CLINICAL TRIAL: NCT04591054
Title: Single-center, Double-arm, Prospective Clinical Trial to Compare Visual Performance of Non-diffractive Extended Vision and Neutral Aspheric Monofocal Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seth M Pantanelli, Associate Professor of Ophthalmology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15524
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cataract; Presbyopia
Keywords: extended vision; intraocular lens; presbyopia; enVista; Vivity
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: single-center, double-arm, patient and assessor blinded
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Extended Vision IOL (Active Comparator): Vivity
  Interventions: Device: Extended Vision IOL
- Neutral Aspheric Monofocal IOL (Active Comparator): enVista [MX60E]
  Interventions: Device: Neutral Aspheric Monofocal IOL

INTERVENTIONS:
Device: Extended Vision IOL — Vivity IOL implantation following cataract extraction
  Arms: Extended Vision IOL
Device: Neutral Aspheric Monofocal IOL — enVista IOL implantation following cataract extraction
  Arms: Neutral Aspheric Monofocal IOL

SUMMARY:
The purpose of this study is to compare the binocular distance, intermediate, and near visual acuity of the Alcon Vivity and Bausch & Lomb enVista IOLs.

We hypothesize that the Alcon Vivity and Bausch & Lomb enVista IOLs will have similar distance, intermediate, and near visual acuity. If the null hypothesis is rejected, then the visual performance of the IOLs may be different.

DETAILED DESCRIPTION:
Presbyopia correcting intraocular lens (PC-IOL) technology has been available for decades. Lens designs have included refractive (e.g. AMO ReZoom), apodized diffractive (e.g. Alcon Acrysof ReSTOR/PanOptix), accommodating (B&L Crystalens), and extended depth-of-focus (e.g. J&J Symfony) technology. Spectacle independence is significantly higher with PC-IOLs when compared with that of monofocal IOLs.1,2 Despite their clear benefits, PC-IOLs are not without drawbacks. Any IOL that splits light to deliver distinct distance and near foci creates the potential for photic phenomenon, which patients may perceive as glare, haloes, and starbursts.3,4

Pseudoaccommodation is defined as an increased depth-of-focus in an emmetropic eye that does not have the ability to change its refractive power. Spherical aberration, which may come from the cornea or IOL, plays an important role in pseudoaccommodation.5,6 There is a small body of literature that IOLs (e.g. Mini WELL, SIFI, Catalina, Italy) with highly-positive spherical aberration can result in significant pseudoaccommodation and lower unwanted optical phenomena than current multifocal IOLs.7

The Alcon Vivity PC-IOL is a hydrophobic acrylic, non-diffractive, extended depth of focus IOL designed for implantation in the capsular bag following cataract extraction. The single-piece IOL has a 6.0 mm diameter and has a hyper-prolate profile that extends the depth of focus to deliver a broader range of sharp vision, with the glare and halo profile approaching that of a monofocal IOL.8

The Bausch & Lomb enVista MX60E is a posterior chamber hydrophobic acrylic IOL. The single-piece IOL has a 6.0 mm diameter and has a neural aspheric optical profile. This neutral aspheric profile, combined with the cornea's natural positive spherical aberration, may extend the depth of focus relative to other negative aspheric hydrophobic acrylic monofocal IOLs on the market.

To date, there is no existing literature comparing the visual performance and patient reported outcomes of the two above mentioned lens technologies; namely, one that relies on a non-diffractive, hyper-prolate profile and another that relies on the cornea's natural positive spherical aberration to provide pseudoaccommodation.

The FDA Summary of Safety and Effectiveness on the Alcon Vivity IOL compares visual and patient reported outcomes of the Alcon Vivity IOL and the Alcon Acrysof SN60WF. While the Alcon Acrysof SN60WF and Bausch & Lomb enVista lenses are not identical, they are considered similar. The document reported improved intermediate vision with the Alcon Vivity over the SN60WF, and rates of reported visual disturbances were similar between the two devices.

Whereas the Alcon Acrysof SN60WF has a negative aspheric optical profile, the Bausch & Lomb enVista has a neutral aspheric optical profile. Theoretically, the Bausch & Lomb enVista IOL may provide increased intermediate vision compared with the SN60WF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 or older at the time of study enrollment.
* Visually significant cataract in the study eyes for which phacoemulsification cataract extraction and posterior chamber IOL implantation is indicated.
* Anticipated to undergo bilateral sequential cataract surgery
* Projected postoperative CDVA 0.20 logMAR (Snellen 20/32) or better in the study eyes, as determined by an Investigator's medical judgement.
* Calculated spherical power targeted at emmetropia at distance in the study eyes.
* Calculated IOL power between +15.0 - +25.0 D, inclusive, in both eyes.
* Measured against-the-rule astigmatism less than 0.6 D or with-the-rule/oblique astigmatism less than 1.25 D.
* If wearing rigid gas permeable (RGP) contact lens in the study eye, willingness to discontinue lens wear for ≥ 21 days prior to preoperative biometry.
* Availability, willingness, and sufficient cognitive awareness to return for study-required visits and comply with examination procedures.
* Willingness to sign the IRB-approved informed consent form (ICF) for study participation.

Exclusion Criteria:

* Mature cataract in the study eye that is likely to prolong surgical procedure and/or lead to intraoperative complications prior to attempted IOL implantation.
* Any visually significant intraocular media opacity other than cataract in the study eye (as determined by the investigator). Such opacities might include corneal scar or vitreous hemorrhage.
* Abnormal corneal findings in the study eye (e.g. keratoconus, pellucid marginal degeneration, irregular astigmatism).
* Any anterior segment pathology in the study eye that could significantly affect outcomes (e.g. chronic uveitis, iritis, aniridia, clinically significant corneal dystrophies, poor pupil dilation, etc.)
* Any condition in the study eye that could affect IOL stability (e.g. pseudoexfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc.).
* History of severe dry eye in the study eye that, in the judgement of the investigator, would impair the ability to obtain reliable study measurements.
* History of serious corneal disease (e.g. herpes simplex, herpes zoster keratitis, etc.) in the study eye.
* History of any clinically significant retinal pathology or ocular diagnosis in the study eye that could, in the investigator's best judgement, alter or limit final post-operative visual prognosis (e.g. diabetic retinopathy, ischemic disease, macular degeneration, retinal detachment, optic neuropathy, amblyopia, strabismus, aniridia, epiretinal membrane, etc.).
* History of cystoid macular edema in either eye.
* History of uveitis in either eye.
* History of intraocular or corneal surgery in the study eye besides laser peripheral iridotomy (LPI), selective laser trabeculoplasty (SLT), or argon laser trabeculoplasty (ALT).
* Uncontrolled glaucoma in the study eye (per Investigator judgement).
* Current ocular infection in the study eye.
* Presence of uncontrolled systemic disease that could increase operative risk (e.g. diabetes mellitus, mental illness, dementia, clinically significant atopic disease, etc.).
* Planned concomitant ocular procedure during cataract surgery inclusive of glaucoma surgery e.g. MIGS or limbal relaxing incisions.
* Symptoms that might be consistent with active COVID-19 including fever, chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches.
* If COVID-19 positive, at least two weeks since last symptoms.
* Unsuitable for study participation for any other reason, as determined by the Investigator's clinical judgement.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center Eye Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Vision IOL | Neutral Aspheric Monofocal IOL
Started | 28 | 28
Completed | 24 | 27
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Vision IOL | Neutral Aspheric Monofocal IOL | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6.3) | 66 (8.1) | 66.5 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 21 | 25 | 46
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Binocular Intermediate Vision
Description: Mean logMAR best-distance corrected visual acuity at intermediate (66 cm) tested in binocular photopic conditions at 3 months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Extended Vision IOL | Neutral Aspheric Monofocal IOL
Number analyzed (Participants) | 24 | 27
logMAR | -0.02 (0.13) | 0.19 (0.14)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Extended Vision IOL | Neutral Aspheric Monofocal IOL
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 3/24 | 5/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Vision IOL (N=24) | Neutral Aspheric Monofocal IOL (N=27)
Cystoid Macular Edema (Eye disorders) | 1 (1) | 1 (1)
Corneal Abrasion (Eye disorders) | 0 (0) | 2 (2)
increased intraocular pressure (Eye disorders) | 1 (1) | 0 (0)
Breakthrough inflammation (Eye disorders) | 1 (1) | 1 (1)
Prolonged corneal edema (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04591054/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT04591054/ICF_001.pdf